CLINICAL TRIAL: NCT03038828
Title: Phase 1 Dose Escalation Study to Establish the Safety of Leukocyte Interleukin, Injection for Treatment of Perianal Warts in Adult Men and Women Who Are HIV/HPV Co-infected
Brief Title: Study of Leukocyte Interleukin, Injection for Treatment of Perianal Warts
Acronym: PAW
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: CEL-SCI Corporation (Industry)
Collaborators: Ergomed Clinical Research Inc. (Unknown); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: NMCSD2013.008_UCSF - deleted
Record Dates: First submitted 2016-09-08; First posted 2017-02-01 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2022-05

CONDITIONS: Perianal Warts
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Cohort A - 200IU Leukocyte Interleukin, Injection 5 days/week x 2 weeks, off two weeks, then repeat 200IU 5 days/week x 2 weeks.
  Interventions: Biological: Leukocyte Interleukin, Injection
- Arm B (Experimental): Arm B - 400IU Leukocyte Interleukin, Injection 5 days/week x 2 weeks, off 2 weeks, 400IU 5 days/week x 2 weeks.
  Interventions: Biological: Leukocyte Interleukin, Injection

INTERVENTIONS:
Biological: Leukocyte Interleukin, Injection — Immunotherapy
  Other Names: Multikine

SUMMARY:
Study is a dose escalation study. Fifteen patients will be enrolled in 2 treatment cohorts. Five participants (cohort A) will be treated with 200IU Multikine daily, 5 days/week for 2 weeks, off 2 weeks, then again 5 days/week for 2 weeks. If no serious adverse events are noted in cohort A patients, ten participants will be treated in cohort B. Cohort B participants will be treated the same as cohort A participants except that dose will be increased to 400IU Multikine per day.

DETAILED DESCRIPTION:
Study is a dose escalation study to determine the safety of Leukocyte Interleukin, Injection in treating men and women with perianal warts who are HIV/HPV co-infected. Fifteen patients will be enrolled in 2 treatment cohorts. Five participants (cohort A) will be treated with 200IU Multikine daily, 5 days/week for 2 weeks, off 2 weeks, then treated again 5 days/week for 2 weeks. If no serious adverse events are noted in cohort A patients, ten (10) participants will be treated in cohort B. Cohort B participants will be treated in the same manner as cohort A participants except that the dose will be increased to 400IU Multikine per day.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Diagnosed with perianal condyloma by primary clinician
3. HIV-infected, may be on or off of antiretroviral therapy. Enrolment of subjects on HAART will be restricted to those individuals for whom an alternative regimen can reasonably be constructed in case of failure.
4. Negative reaction to intradermal test with ciprofloxacin (a fluoroquinolone antibiotic)
5. Any CD4 count will be considered appropriate for study
6. Blood WBC > 2.0x103/mm3 and absolute neutrophils count > 500
7. Blood hemoglobin > 10.0 g/dL
8. Blood platelet count > 50x103/mm3
9. Serum total bilirubin < 6.0 mg/dL (participants taking atazanavir-based ARV regimens may have elevated total bilirubin but are generally < 6)
10. Blood aspartate aminotransferase (AST) < 100 U/L (<2 ULN)
11. Blood alanine aminotransferase (ALT) < 130 U/L (<2 ULN)
12. Serum creatinine < 1.5 mg/dL
13. ECOG performance status < 3
14. If a subject is of reproductive potential he/she and her/his sexual partner MUST be willing and able to utilize highly effective methods of contraception (e.g., birth control pill, barrier methods with spermicide - as applicable) for the duration of the study including the study follow-up period.
15. Subjects must be willing to refrain from anal sex, douching and use of enemas prior to scheduled Pap smears

Exclusion Criteria:

1. Anal cancer (current or history of)
2. Inability to attend study visits
3. Participation in any other drug study
4. History of asthma
5. History of CHF and/or cardiac support for arrhythmia or on chronic cardiac medication or has other chronic or acute cardiac ailments (e.g., or abnormal EKG at Baseline)
6. History of organ transplantation or requiring chronic administration of immune suppressive drugs in the last 6 months
7. For women, neither pregnant nor lactating
8. In the opinion of the Primary Investigator, the subject may not be able to tolerate the study treatment regimen
9. Subjects who are currently using or have recently within past 3 months) been treated with immunomodulators (e.g., Interferon-α)
10. Subjects with active infections including sexually transmitted diseases (e.g., N. gonorrhea, C. trachomatis, H. ducreyi, T. pallidum)
11. History of allergic reaction to fluoroquinolone antibiotics (e.g., ciprofloxacin, ofloxacin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Wart characterization change | Time Frame: Days 0, 4, 11, 32, 39, 70, 100, 130, 160 ]
  Perianal wart characterization includes counting the number of identified warts, the diameter measurement of each identified wart in millimeters and the photographic imaging of each identified wart during the treatment phase and the follow-up phase of the study

SECONDARY OUTCOMES:
Assessment of HPV subtype identification change | Days 0, 4, 11, 32, 39, 70, 100 130, 160
  HPV subtyping will be performed on specimens collected from the anal canal.
Assessment of Anal dysplasia cytologic grade change | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  Anal dysplasia cytologic specimen collection will take place during the treatment phase and the follow-up phase of the study
Assessment of adverse effects during the treatment phase of the study assessed | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  Adverse effects experienced during the treatment phase of the study are recorded by the study participants in a symptoms log

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Talor, PhD, Study Director — CEL-SCI Chief Scientific Officer
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No